CLINICAL TRIAL: NCT01675830
Title: Heat Retention Head Wrap Use for Re-warming of Infants Requiring Cardio-Pulmonary Bypass
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cardiology Clinical Research & Regulatory Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-P00001161
Record Dates: First submitted 2012-07-19; First posted 2012-08-30 (Estimated); Results first posted 2015-02-26 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Impaired Thermoregulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Head Retention Head Wrap device (Experimental): All subjects recieved the experimental intervention with the Heat Retention Head Wrap device for during the rewarming phase of cardiopulmonary bypass surgery.
  Interventions: Device: Heat Retention Head Wrap

INTERVENTIONS:
Device: Heat Retention Head Wrap — Applied to infant's heads during the rewarming phase of CBP surgery

SUMMARY:
This is a phase I descriptive pilot study to determine the feasibility of using the Heat Retention Head Wrap on infants during the re-warming period following cardio-pulmonary bypass.

DETAILED DESCRIPTION:
According to the World Health Organization a body temperature of 36-36.5 degrees Celsius is mild hypothermia, 32-36 degrees Celsius is moderate hypothermia, and < 32 degrees Celsius is severe hypothermia.1 Hypothermia can be a major postoperative problem for infants undergoing cardio-pulmonary bypass (CPB) surgery. During CPB, patients are cooled to decrease metabolism and protect myocardium and brain. When the repair is completed, the patient is re-warmed as the temperature of blood in the bypass pump is gradually increased. However, after separation from the CBP pump, infants consistently experience a temperature drop of 2 to 5 degrees Celsius.

With head cooling heat dissipates more quickly than with any other body surface. As much as 60% of an infant's body heat can dissipate through an uncovered head, thus leaving patients at high risk for complications associated with hypothermia. The amount of heat lost to the environment by newborn infants has a great impact on mortality rates, growth, and energy maintenance. Major adverse effects from inadvertent hypothermia include myocardial ischemia, impaired coagulation, prolonged healing, surgical wound infections, and decreased postoperative comfort.

Nursing participation in the re-warming of patients during CPB surgery is a core intervention. According to recommendations for perioperative registered nurses the patient should be at or returning to normothermia at the conclusion of the immediate postoperative period. Current standards of care for re-warming after CPB do not include any particular type of head covering. Recently, a new head covering made of biaxial-oriented polyethylene terephthalate (boPET), called the Heat Retention Head Wrap, has been designed for use with infants to facilitate warming during the postoperative period (that begins during the re-warming phase of CBP). The purpose of this study will be to determine the feasibility of using the Heat Retention Head Wrap on infants during the re-warming period following CPB.

Specific Aims

1. To describe the feasibility of placing a Heat Retention Head Wrap on the infant's head from the time the re-warming process begins to the time baby arrives in the Cardiac Intensive Care Unit (CICU) after transfer from the operating room.
2. To characterize the temperature progression from (1) the onset of re-warming, (2) removal of bypass cannulas, to (3) removal of the rectal temperature probe immediately before transfer from the OR to the CICU, and (4) upon arrival to the CICU.
3. To identify and describe adverse events observed with use of the Heat Retention Head Wrap.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing CPB surgery.
* Weigh ≥ 3 and ≤ 10 kg.
* Cooled to 24-30 degrees Celsius.
* Head circumferences between 33-48 cm.
* Scalp free of skin lesions such as reddened areas, ulcerations, abrasions, burns, and hemangiomas.

Exclusion Criteria:

* Require cooling below 24 degrees Celsius at any point during CPB surgery.
* Weigh less than 3 kg or more than that 10kg.
* Are premature or < 37 weeks corrected gestational age.
* Have a head circumference smaller than 33 cm or larger than 48 cm.
* Have a known or previously diagnosed neurological trauma, malignant hyperthermia, stroke, seizure, VP shunt, evidence of scalp lesions, or other known comorbidity.
* Have hair braided close to the scalp.
* Infants with known allergy or sensitivity to polyethylene terephthalate (known as Mylar)

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2011-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Sakakeeny, BSN, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Head Wrap Device: Heat Retention Head Wrap: Applied to infant's heads during the rewarming process of CPB
Period: Overall Study
Arm/Group | Head Wrap Device
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Head Wrap Device
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: weeks] | 17.4 [4.3 to 47.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Head Wrap Feasibility
Description: To describe the feasibility of placing a Thermoregulation Head Wrap on the infant's head from the time the re-warming process begins to the time baby arrives in the Cardiac Intensive Care Unit (CICU) after transfer from the operating room. Likert scale items assessing feasibility of the head wrap will be completed by clinicians upon patient admission to CICU.
Time Frame: <12 hours
Population: Percentage of respondents that agree device is easy to use
Measure: Number; unit: percentage of respondents
Arm/Group | Head Wrap Device
Number analyzed (Participants) | 10
percentage of respondents | 100

2. Secondary Outcome: Redness, Irritation, and/or Hyperthermia Due to Head Wrap Use
Description: To identify and describe adverse events observed with use of the Thermoregulation Head Wrap.
Time Frame: These will be assessed upon admission to the CICU, and in 6 hour follow up increments until the last assessment at 72 hours.
Population: Number of adverse events observed
Measure: Number; unit: adverse events
Arm/Group | Head Wrap Device
Number analyzed (Participants) | 10
adverse events | 0

ADVERSE EVENTS:
Time Frame: 72 hours following application of the head wrap device
Arm/Group | Head Wrap Device
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
Investigators could not account for differences in the room temperature, heated and humidified gases, CPB regulation, regulation of forced air warming system, warming of IV fluids, and temperature of irrigation solutions in the OR.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No